CLINICAL TRIAL: NCT03240185
Title: Effectiveness of Guided Breathing Exercises on Anorectal Pain in Patients With Symptomatic Hemorrhoids
Brief Title: Post Hemorrhoidectomy Anorectal Pain
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-36206
Record Dates: First submitted 2017-07-20; First posted 2017-08-07 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Hemorrhoid Pain
Keywords: hemorrhoid; pain; deep breathing; multimodal pain control
MeSH Terms: conditions — Hemorrhoids; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemroidectomy patients: Patients undergoing hemorrhoid surgery who receive education regarding deep breathing exercises for pain control as part of their preoperative appointment
  Interventions: Behavioral: deep breathing exercises

INTERVENTIONS:
Behavioral: deep breathing exercises — Patients receive education on deep breathing exercises for pain control as part of their pre-operative appointment

SUMMARY:
This is a quality assurance trial to evaluate the effectiveness of guided breathing exercises on reducing the symptoms of hemorrhoidal disease in colorectal surgery patients. All patients who undergo hemorrhoid surgery are educated on breathing exercises that can be used to reduce pain and increase relaxation. These patients will be surveyed at their post-operative visit regarding pain and other symptoms and at their one month post operative visit on the any hospitalizations and emergency room visits since their surgery.

DETAILED DESCRIPTION:
The effectiveness of guided breathing exercises on reducing the symptoms of hemorrhoidal disease in colorectal surgery patients will be assessed in this quality assurance trial. During the pre-operative clinic visit, patients to undergo hemorrhoid surgery are educated on breathing exercises that can be used to reduce pain and increase relaxation. In this year long study patient self-reported utilization of the breathing exercises and their level of pain, sleep quality, gastrointestinal symptoms (diarrhea, constipation, etc), emergency room visits, and hospitalizations in the month post hemorrhoid surgery will be evaluated. All patients will be asked to complete a brief survey at their pre-operative and one month post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective hemorrhoid surgery

Exclusion Criteria:

* Emergent/urgent hemorrhoid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in colorectal surgery clinic with planed hemorrhoid surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Pain scores | within ~30 days of surgery, at the time of post-operative clinic visit
  The Wong-Baker faces pain score scale which displays 6 faces with scores of 0, 2, 4, 6, 8, 10, where 0=no hurt and 10=worst hurt will be used in the pre-operative and post-operative surveys to assess each patient's self reported pain level. the lower the score the more favorable/less pain.
Utilization of breathing exercises | within ~30 days of surgery, at the time of post-operative clinic visit
  Response to two questions in the post-operative survey will be used to assess wehether the patient did the breathing exercises after surgery (yes or no) and if they did how man times daily did they do the breathing exercises- <2, 3-5, or >5.

SECONDARY OUTCOMES:
Admissions within 30 Days of Surgery | within 30 days of surgery
  The number of patients who required admission for pain control/infection/bleeding/other complication within 30 days of surgery will be determined from a review of the medical records.
Emergency Department visits within 30 Days of Surgery | within 30 days of surgery
  Evaluating number of patients who visited the Emergency Department within 30 days of surgery will be determined from a review of the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hall, MD, Study Chair — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No